CLINICAL TRIAL: NCT01194518
Title: Exploring Life Experience and Lifestyle Intervention Program Among Patients
Brief Title: Exploring Life Experience and Lifestyle Intervention Program Among Patients With Chronic Kidney Disease: A Longitudinal Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cheng Kung University (Other)
Collaborators: National Cheng-Kung University Hospital (Other); E-DA Hospital (Other)
Responsible Party: Miaofen Yen, National Cheng Kung University
Purpose: Prevention
Other Study IDs: NSC992314B006048MY3
Record Dates: First submitted 2010-08-31; First posted 2010-09-03 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Kidney Disease
Keywords: Life experience; Life style; Health behavior; Mixed method
MeSH Terms: conditions — Renal Insufficiency, Chronic; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle Intervention Program (Experimental)
  Interventions: Behavioral: Lifestyle Intervention Program

INTERVENTIONS:
Behavioral: Lifestyle Intervention Program

SUMMARY:
The lifestyle consulting program through one year follow-up could effective increase the scores of health responsibility and nutrition according to the past three-year study. Behavior change is a dynamic and complex process. Using a long-term follow up approach will be able to understand the trajectory of behavior change. The purpose of this study is to explore life experience and lifestyle intervention program for patients with chronic kidney disease using mixed methods with a longitudinal approach. The first year of this study will include a qualitative study with in depth interview of the subjects who attend previous study in the research team and have the scores of health promoting lifestyle among the highest 27% and lowest 27%. The life experience will be explored. The quantitative study will be an experimental design. Qualified subjects will be randomly assigned to intervention or control group. The intervention protocol is based on trans-theoretical model. Each subject will be followed every six months. The second and third year of studies will continue to use the qualitative and quantitative approach to understand the life experience and meaning among patients with chronic kidney diseases. The trajectory of life experience and life style changes will be explored. The method may strengthen the effectiveness of lifestyle program and may provide comprehensive understanding of the trajectory of behavior changes among patient with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Early Stages of Chronic Kidney Disease (GFR≧30ml/min/1.73㎡)
* Must be able to commmunicate in Chinese or Taiwanese
* Muse be voluntarily to attend
* Patient who does not exercise regularly
* Patient whose blood pressure higher than 140/90 mmHg
* Patient who is overweight or BMI>25kg/㎡

Exclusion Criteria:

* Patient who limited to exercise

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2010-08; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Body weight | six months
Waist to hip ratio | six months
Overall knowledge of renal protection | six months
  The 20 item Renal Protection Knowledge Checklist was developed by researchers will use to measure three dimensions of knowledge: renal function protection, use of Chinese herbs and diet.
Health promotion lifestyle | six months
  Health promotion was measured by 52 item health promotion lifestyle profileⅡ ( HPLP-II).
Quality of Life | six months
  The study will use WHOQOL-BREF to measure the outcome.
Physical activity | six months
  The study will use International Physical Activity Questionnaire (IPAQ) Taiwan version to measure the outcome.
General Health Perceptions | six months
  The study will use General Health Perceptions Subscale of SF-36 Health Status Scale to measure the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan